CLINICAL TRIAL: NCT04250909
Title: Retrospective 5-year Safety Analysis of the BIOLUX P-I and P-II Studies in Subjects Requiring Revascularization of Infrainguinal Arteries
Brief Title: Retrospective Follow-up of BIOLUX P-I/-II
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1901
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Overall Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passeo 18 PTA: Previous treatment with uncoated Passeo 18 PTA balloon catheter
  Interventions: Device: Passeo-18
- Passeo-18 Lux DCB: Previous teatment with Passeo-18 Lux DCB
  Interventions: Device: Passeo-18 Lux

INTERVENTIONS:
Device: Passeo-18 — POBA
  Groups: Passeo 18 PTA
Device: Passeo-18 Lux — DCB
  Groups: Passeo-18 Lux DCB

SUMMARY:
The aim is to collect long-term clinical data from 132 patients from Belgium, Germany and Austria who had previously participated in either of the BIOLUX P-I or P-II studies. Patients in these studies were treated with either a percutaneous transluminal angioplasty (PTA) balloon catheter or a drug-coated Passe-18-Lux balloon (DCB). The purpose of Retro-BIOLUX P-I-II is to collect clinical data from patients treated with either Passeo-18 PTA or Passeo-18 Lux DCB to analyze the long-term effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was previously enrolled in either BIOLUX P-I or BIOLUX P-II
2. Subject was treated either with Passeo-18 PTA or Passeo-18 LUX
3. Written informed consent by subject or subject's legal representative or impartial witness/waiver

Exclusion Criteria:

1. Subject did neither participate in BIOLUX P-I nor BIOLUX P-II
2. Subject was neither treated with Passeo-18 Lux nor with Passeo-18 PTA
3. Subject is not willing to sign an informed consent /data release form

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from previous studies.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 60 months
  Overall survival at five years after index procedure, defined as death from any cause

SECONDARY OUTCOMES:
Overall survival, defined as the time in days after index procedure to date of death from any cause. | 60 months
Major amputations of target extremities | 60 months
Clinically-driven target lesion revascularization | 60 months
Cause of death (descriptive analysis) at five years after treatment within BIOLUX P-I/-II. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof Dr, Study Chair — Clinic of Cardiology and Angiology II Bad Krozingen
Locations (8):
- Austria (2):
  - LKH Univ.-Klinikum Graz, Ambulanz für Angiologie, Graz
  - Allgemeines Krankenhaus - Universitätsklinik für Radiodiagnostik, Klinische Abteilung für Kardiovaskuläre und Interventionelle Radiologie, Vienna
- Belgium (2):
  - Vascular Research Center Bornheiden, Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
- Germany (4):
  - Clinic of Cardiology and Angiology II Bad Krozingen, Bad Krozingen
  - Gefäßzentrum am KEH, Berlin
  - University Leipzig Medical Centre Medizinische Klinik und Poliklinik V (Angiologie), Leipzig
  - Institut für Diagnostische und Interventionelle Radiologie, RoMed Klinikum, Rosenheim